CLINICAL TRIAL: NCT06174935
Title: Low Dose Atropine For Symptomatic Vitreous Floaters
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jeanette Du (Other)
Responsible Party: Sponsor-Investigator, Jeanette Du, Physician, Prism Vision Group
Organization: Prism Vision Group (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1362664
Record Dates: First submitted 2023-11-28; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Vitreous Floaters
MeSH Terms: conditions — vitreous floaters

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Atropine 0.01% (Experimental): Patients will apply 1 drop daily of atropine 0.01%
  Interventions: Drug: 0.01% atropine ophthalmic drop

INTERVENTIONS:
Drug: 0.01% atropine ophthalmic drop — 0.01% atropine ophthalmic drop will be applied daily to the affected eye

SUMMARY:
The objective of this study is to identify a potential pharmacologic option by assessing whether 0.01% atropine may be effective for treating bothersome floaters as measured by scores on a modified NEI VFQ-25.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients within Prism Vision Group with ICD diagnosis of acute posterior vitreous detachment and none of the ocular comorbidities listed as exclusion criteria will be screened as potential study participants.

Exclusion Criteria:

* Patients with vitreous hemorrhage, other significant media opacity or vitreoretinal pathology, or history of pars plana vitrectomy will be excluded.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Symptom improvement assessed by questionnaire | Up to 2 months
  NEI VFQ-25 = National Eye Institute Visual Function Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Retina Group of Washington, Reston, Virginia, United States

IPD SHARING:
Plan to Share IPD: No